CLINICAL TRIAL: NCT00002015
Title: An Open Label Evaluation of the Safety and Pharmacokinetics of Ganciclovir in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roche Global Development (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 029G; ICM 1788
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; Ganciclovir; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Immunocompromised Host
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
To evaluate the pharmacokinetics of intravenous ganciclovir in children (ages 3 months - 12 years). To determine the safety and tolerance of a 2 to 3 week induction course of ganciclovir IV in immunocompromised children receiving treatment for life- or sight-threatening cytomegalovirus infections.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Topical acyclovir.
* Consult with the Syntex study monitor for the following:
* Cytokines.
* Soluble CD4.
* Trichosanthin (Compound Q).
* Imipenem-cilastatin.
* Other investigational drugs.

Patients must have the following:

* Congenital or acquired immune deficiency.
* Eligibility to receive ganciclovir for the treatment of life- or sight-threatening Cytomegalovirus (CMV) disease.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Mild to moderate Cytomegalovirus infection that does not satisfy the clinical severity criteria.
* Congenital or neonatal CMV infections without documented congenital or acquired immunodeficiency.

Concurrent Medication:

Excluded:

* Other myelosuppressive drugs.
* Antimetabolites.
* Alkylating agents.
* Nucleoside analogs (topical acyclovir is allowed).
* Interferons.
* Foscarnet.
* Consult with the Syntex study monitor for the following:
* Cytokines.
* Soluble CD4.
* Trichosanthin (Compound Q).
* Imipenem-cilastatin.
* Other investigational drugs.

Patients with the following are excluded:

* Mild to moderate Cytomegalovirus (CMV) infection that does not meet the clinical severity criteria.
* Absolute neutrophil count (ANC) < 500 cells/mm3 or a platelet count < 25000 platelets/mm3. Note:
* Exceptions may be made for patients with pre-existing neutropenia or thrombocytopenia and immediately life-threatening disease, if the investigator believes that a delay in starting ganciclovir therapy is not advisable. In such patients, the investigator should advise the parents or guardians of the risk of further bone marrow suppression and the increased risk of infection or bleeding.
* Receiving excluded medications that it is not possible to discontinue.
* Congenital or neonatal CMV infections without documented congenital or acquired immunodeficiency.
* Demonstrated hypersensitivity to acyclovir or ganciclovir.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hosp of Los Angeles, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Ctr for the Health Sciences / UCLA Med Ctr, Los Angeles, California
  - Univ of Chicago / Wylers, Chicago, Illinois
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - Univ of Rochester Med Ctr, Rochester, New York
  - Baylor College of Medicine / Texas Children's Hosp, Houston, Texas